CLINICAL TRIAL: NCT00587327
Title: A Randomised, Double-blind, Parallel Groups, Placebo-controlled, Multi-centre Study Assessing the Effects of a Selective Oxytocin Antagonist (Barusiban) and a Mixed Oxytocin Antagonist - Vasopressin V1a Antagonist (Atosiban) Administered Intravenously on Luteal Phase Uterine Contractions in Oocyte Donors Supplemented With Vaginal Progesterone
Brief Title: Effect of Oxytocin and Vasopressin Antagonists on Uterine Contractions
Acronym: OVANCON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FE200440 CS09
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: In Vitro Fertilisation (IVF) Treatment
MeSH Terms: interventions — barusiban; atosiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Barusiban (Experimental)
  Interventions: Drug: Barusiban
- Atosiban (Experimental)
  Interventions: Drug: Atosiban
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Barusiban — Solution for IV treatment. Bolus and infusion for 4 hours
  Arms: Barusiban
Drug: Atosiban — Solution for IV administration. Bolus and infusion for 4 hours
  Arms: Atosiban
Drug: Placebo — Saline solution for IV administration. Bolus and infusion for 4 hours.
  Arms: Placebo

SUMMARY:
The main purpose of this clinical research trial was to evaluate the effects of barusiban and atosiban compared to placebo on luteal phase uterine contractions in oocyte donors supplemented with progesterone.

DETAILED DESCRIPTION:
This was a randomised, double-blind, parallel groups, placebo-controlled, multi-centre trial. It was designed to evaluate the effects of a selective oxytocin antagonist (barusiban) and a mixed oxytocin antagonist - vasopressin V1a antagonist (atosiban) on uterine contractions during the luteal phase. Participants in this trial were oocyte donors who had undergone controlled ovarian hyperstimulation in the long gonadotrophin-releasing hormone (GnRH) agonist protocol or the multiple-dose or single-dose GnRH antagonist protocols, received hCG for triggering of final follicular maturation and undergone oocyte retrieval (OR). The duration of the trial was five days and participants attended the clinic on three occasions: Day OR +1 (screening), Day OR +2 (randomisation and dosing of investigational medicinal product), and Day OR +5 (end-of-trial).

After screening on Day OR +1, participants initiated luteal support supplementation with vaginal progesterone, which continued throughout the trial. On Day OR +2, participants were randomised to either barusiban, atosiban or placebo and participants received an intravenous (IV) bolus followed by an IV infusion of either barusiban, atosiban or placebo for approximately 4h. A mock embryo transfer was performed 3h after start of dosing.

Uterine contractility parameters were assessed by transvaginal ultrasound. The transvaginal ultrasound recordings were analysed for uterine contractions by a central independent assessor, blinded to treatment allocation

Definitions:

The frequency of uterine contractions was defined as the number of uterine contractions per minute. A contraction was defined as one sequential upward and downward vertical displacement of the endometrial / myometrial interface over time.

The external contractile measure was the mean wave amplitude in mm at the lumenal surface. This metric was measured at the lumenal peaks and troughs only and was a measurement designed to study the relationship between endometrial wave activity, manifested as bulk motion of the uterus, versus internal contractile strength. The external contractile measure was reported in mm/contraction.The external contractile measure quantified the movement of the uterus as a whole as measured at the lumen, i.e. the motion of the uterus relative to the body.

The internal contractile measure was the strength of the contractions based upon the sum of the contraction amplitudes measured at the anterior and posterior endometrial / myometrial interfaces. The amplitude at each interface was defined as the average difference between the endometrial / myometrial-lumenal distance measured at the peaks and troughs of the endometrial / myometrial interfaces. The internal contractile measure was reported in mm/contraction. The internal contractile measure quantified the movement of the endometrium relative to the lumen, i.e. the motion internal to the uterus.

The total contractile measure was the sum of the external contractile measure and the internal contractile measure and quantified total muscle movement in the uterus. If the waves at the anterior and posterior endometrial / myometrial interfaces were in phase then there was no endometrial motion relative to the lumen and the motion was a pure wave motion with the internal contractile measure equal to zero. The total contractile measure was reported in mm/contraction.

Inter-subendometrial space was measured as the distance between the anterior stratum basalis and posterior stratum basalis layers in mid-sagittal plane at an anatomic location between 5 and 10 mm from the fundus. All inter-subendometrial space measurements were made by selecting a clear image of the uterus, waiting for any contractions to pass and freezing the image.

A linear distance measurement was then taken between the anatomic landmarks described above. Inter-subendometrial space was calculated from existing measurements using the mean of all measurements identifying the endometrial-myometrial interfaces on the superior and inferior surfaces in each endometrial strip when the arrows identifying endometrial contractions were placed for motion analysis. Inter-subendometrial space was reported in mm

ELIGIBILITY:
Participants eligible for this trial were oocyte donors 18-35 years of age, who had undergone controlled ovarian hyperstimulation in the long GnRH agonist protocol or the multiple-dose or single-dose GnRH antagonist protocols, had received hCG (≥ 5,000 IU urinary hCG or 250 μg recombinant hCG) for triggering of final follicular maturation and had undergone oocyte retrieval with a yield of ≥ 6 cumulus-oocyte-complexes. Participants had given signed informed consent, were generally healthy and with a body mass index (BMI) of 18.5-29.9 kg/m2. Participants were excluded in case of endometriosis stage I-IV or uterine pathology. Participants were willing to not have intake of alcoholic beverages during the trial, to not have sexual intercourse during the trial, and to either maintain sexual abstinence or use a highly effective method of contraception from end-of-trial till onset of next menses.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Frequency of uterine contractions | 3h after start of dosing

SECONDARY OUTCOMES:
Period, external contractile measure, internal contractile measure and total contractile measure of uterine contractions | 3h after start of dosing
Frequency, period, external contractile measure, internal contractile measure and total contractile measure of uterine contractions | 5 min, 15 min, 30 min, 1h, 1h 30 min, 2h, and 2h 30 min after start of dosing
Frequency, period, external contractile measure, internal contractile measure and total contractile measure of uterine contractions | 5 min, 30 min, and 1h after mock embryo transfer
Frequency, period, external contractile measure, internal contractile measure and total contractile measure of uterine contractions | 30 min and 1h post-dosing and on Day OR +5
Inter-subendometrial space | 5 min, 15 min, 30 min, 1h, 1h 30 min, 2h, 2h 30 min, and 3h after start of dosing, at 5 min, 30 min, and 1h after mock embryo transfer, at 30 min and 1h post-dosing and on Day OR +5
Pharmacokinetic parameters of barusiban and atosiban | 2 days after oocyte retrieval (Day OR +2, sampling throughout the day) and 5 days after oocyte retrieval (Day OR +5, one sampling)
Population pharmacokinetic / pharmacodynamic model | 30 min and 3h after start of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (5):
- UZ Brussel, Center for Reproductive Medicine, Brussels, Belgium
- Czechia (2):
  - Institute for Reproductive Medicine and Endocrinology, Pilsen
  - ISCARE IVF a.s., Prague
- Spain (2):
  - Institut Universitari Dexeus, Barcelona
  - IVI Madrid, Madrid